CLINICAL TRIAL: NCT01069913
Title: A Pharmacokinetics Profile Determination of BG00012 Standard Formulation and the BG00012 Active Pharmaceutical Ingredient (API) After a Single Oral Dose Administered to Healthy Male Volunteers
Brief Title: Pharmacokinetics Profile Study of BG00012 Standard Formulation and BG00012 Active Pharmaceutical Ingredient
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec, Medical Director
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 109HV105
Record Dates: First submitted 2010-02-12; First posted 2010-02-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: Healthy Volunteer
MeSH Terms: interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BG00012 (Active Comparator): BG00012 Standard Formulation
  Interventions: Drug: BG00012
- BG00012 API (Active Comparator): BG00012 API
  Interventions: Drug: BG00012

INTERVENTIONS:
Drug: BG00012 — Sequence 1: Oral 240 mg BG00012 Standard Formulation & Following 7 day washout period, 240 mg BG00012 API.
  Sequence 2: 240 mg BG00012 API & Following 7 day washout period, 240 mg BG00012 Standard Formulation.

SUMMARY:
The purpose of this study is to measure two different formulations of BG00012 to determine how much of each formulation of BG00012 reaches the blood stream and how long it takes the body to get rid of it, when given as a single dose.

ELIGIBILITY:
Inclusion Criteria:

1. Males 18 to 55 years old, inclusive, at the time of informed consent.
2. Must weigh between 50 kg and 110 kg, inclusive.
3. Must have a body mass index (BMI) between 19 kg/m2 and 30 kg/m2, inclusive.
4. All subjects must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.
5. Must be a non-smoker, and no use of chewing tobacco, for at least 6 months prior to Day -1.
6. Must have a screening physical examination and ECG without any clinically significant abnormality (as determined by the Investigator).

Exclusion Criteria:

1. History of malignancy (subjects with basal cell carcinoma that has been completely excised prior to study entry remain eligible).
2. History of severe allergic or anaphylactic reaction.
3. History of any clinically significant endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major diseases, as determined by the Investigator.
4. Clinically significant abnormal hematology or blood chemistry values, as determined by the Investigator.
5. Serious infection (e.g., pneumonia, septicemia) within the 2 months prior to Day -1.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
PK profiles of the current BG00012 standard formulation and the BG00012 API formulation in healthy volunteers. Primary PK parameter will be the area under the plasma concentration curve | 4 days post dosing period 2

SECONDARY OUTCOMES:
To assess the safety and tolerability of the current oral BG00012 standard formulation and the encapsulated oral BG00012 API | 4 days after dosing period 2

CONTACTS AND LOCATIONS:
Overall Officials: Biogen Idec Medical Director, Study Director — Biogen Idec, Cambridge, MA USA